CLINICAL TRIAL: NCT03342911
Title: Nivolumab Plus Weekly Carboplatin and Paclitaxel as Induction in Resectable Locally Advanced Head and Neck Cancer
Brief Title: Nivolumab, Carboplatin, and Paclitaxel in Treating Patients With Stage III-IV Head and Neck Squamous Cell Carcinoma That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.513; JT 11182 (Other: JeffTrial Number)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Name Human Papillomavirus Positive Oropharyngeal Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma; Stage III Laryngeal Squamous Cell Carcinoma; Stage III Oral Cavity Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IV Laryngeal Squamous Cell Carcinoma; Stage IV Oral Cavity Squamous Cell Carcinoma; Stage IV Oropharyngeal Squamous Cell Carcinoma; Stage IVA Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Hypopharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Oral Cavity Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Hypopharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Oral Cavity Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; Taxes; Carboplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, paclitaxel, carboplatin) (Experimental): Patients receive nivolumab IV over at least 30 minutes on day 1, paclitaxel IV on days 1 and 8, and carboplatin IV on days 1 and 8. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Nivolumab

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: 125973; 33069-62-4; 673089; Anzatax; Asotax; Bristaxol; Taxol; Praxel
Drug: Carboplatin — Given IV
  Other Names: Carboplat; Carboplatin Hexal; Ribocarbo; Carbosol
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; ONO-4538

SUMMARY:
This phase II trial studies how well nivolumab, carboplatin, and paclitaxel work in treating patients with stage III-IV head and neck squamous cell carcinoma that can be removed by surgery. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab, carboplatin, and paclitaxel may work better in treating patients with head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate pathologic complete response (pCR) at the primary site in patients with newly diagnosed and untreated stage III-IVA squamous cell carcinoma of the head and neck (SCCHN) of the oral cavity, oropharynx, larynx, and hypopharynx with nivolumab, paclitaxel and carboplatin in addition to standard chemotherapy.

SECONDARY OBJECTIVES:

I. Safety. II. Complete pathologic response at all sites of disease. III. Major pathologic response rate at primary site. IV. Overall clinical response rate. V. Clinical complete response rate. VI. 1 year progression-free survival (PFS). VII. Overall survival.

TERTIARY OBJECTIVES:

I. To explore whether PDL1 expression is associated with treatment response. II. To explore whether there is a net change in the Th1/Th2 ratio (IFN-gamma, IL-4, IL10, etc.) or cell subset frequencies (M2 monocytes, myeloid-derived suppressor cells, etc.) within a patient's peripheral blood either at baseline or in response to treatment is associated with treatment response.

III. To explore whether exosomes or other immune related serum biomarkers change after combination therapy.

IV. To explore the predictive value of serial cell free deoxyribonucleic acid (DNA) levels and response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age and older.
* Pathologically confirmed SCCHN, not previously treated, with a plan to undergo surgery
* Patients who have stage III-IV disease without distant metastases (M0) of 1) oral cavity, 2) larynx, 3) hypopharynx 4) oropharynx (human papillomavirus [HPV] neg) using American Joint Committee on Cancer (AJCC) 8th edition
* Patients who have oropharyngeal cancer that HPV positive, stage II-III disease without distant metastases (M0) using AJCC 8th edition
* All patients with oropharyngeal SCCHN must be tested for HPV (by p16 and/or HPV in situ hybridization [ISH] or polymerase chain reaction [PCR])
* Patients must be evaluated by a head and neck surgeon and be deemed surgically resectable at baseline
* Tumor sample must be available for HPV p16 and PD-L1 testing and if oropharyngeal, must be tested for HPV p16
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* While blood cells 2000/ul or more
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more; (transfusion permitted)
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x the upper limit of normal
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or serum creatinine less than or equal to 1.5 x upper limit of normal (ULN)
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 21 days of study enrollment
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 23 weeks after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 31 weeks after the last dose of study drugs; men who are azoospermic do not require contraception
* All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Primary nasopharyngeal carcinoma
* Patients who have participated in a study with an investigational agent or device within 2 weeks of initiation of treatment
* Any prior radiotherapy to the neck
* Any prior treatment for SCCHN
* Any prior therapy with anti-PD-1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Any history of a sever hypersensitivity reaction to any monoclonal antibody
* Any history of allergy to the study drug components
* Any concurrent malignancies- exceptions include- basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy; patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post-diagnosis
* Any diagnosis of immunodeficiency or current immunosuppressive therapy including >10mg/day of prednisone within 14 days of enrollment is not permitted (excludes emergency transient steroid use at discretion of the treating physician).
* Patients that have an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (> 10 mg daily prednisone equivalents) or immunosuppressive agents. Subjects with vitiligo, type I diabetes mellitus, or resolved childhood asthma/atopy would be an exception to this rule. Inhaled or topical steroids, and adrenal replacement steroid doses ≤10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Patients with a known human immunodeficiency virus infection (HIV 1/2 antibodies) or acquired immunodeficiency syndrome (HIV/AIDS), active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Patients with evidence of non-infectious pneumonitis or history of interstitial lung disease
* Patients who have received a live vaccine within 30 days prior initiation of the systemic regimen
* Patients must not be receiving any other investigational agents
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial
* Women must not be pregnant (as above) or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (3):
- United States (3):
  - Abington- Jefferson Health, Abington, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Paclitaxel, Carboplatin)
Started | 34
Completed | 30
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: The primary objective of the study is to estimate the rate of pathologic complete response (pCR) at the primary site, defined as the absence of any residual invasive cancer on H&E evaluation of the resected specimen and all sampled ipsilateral lymph nodes, in patients with newly diagnosed and untreated Stage III-IVA SCCHN of the oral cavity, Oropharynx, Larynx, and Hypopharynx treated with standard neoadjuvant chemotherapy plus Nivolumab, paclitaxel, and carboplatin. Pathologic complete response rate and its associated score 95% confidence interval will be estimated.
Time Frame: Up to 26 months
Population: The complete pathologic response rate was 45.45% (15/33) with a 95% Confidence Interval of 28.5% to 63.4%.
Measure: Number (95% Confidence Interval); unit: percentage of complete response
Arm/Group | Treatment (Nivolumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 33
percentage of complete response | 45.5 [28.5 to 63.4]

2. Secondary Outcome: Number of Patients Who Achieved Major Pathologic Response (Defined as 10% or Less Residual Viable Tumor)
Description: patients achieved the major pathologic response (i.e., <10% viable tumor) or pathologic complete response
Time Frame: Up to 26 months
Population: number of patients with Major response (Major or complete) was 72.73% (24/33) with a 95% Confidence Interval of 54.2% to 86.1%.
Measure: Number (95% Confidence Interval); unit: percentage of major response
Arm/Group | Treatment (Nivolumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 33
percentage of major response | 72.73 [54.2 to 86.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected starting Day 1 of study treatment, and continue for up to 100 days after the last study treatment (Day 156 +/- 5 days) or last day of study participation (up to Day 156 +/- 5 days). At each study visit, the investigator (or designee) will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization for approximately 6 months.
Description: An adverse event is any untoward or unfavorable medical occurrence in a human participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Treatment (Nivolumab, Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 5/34
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Paclitaxel, Carboplatin) (N=34)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
low absolute neutrophil count grade 4 (Blood and lymphatic system disorders) | 2 (2)
Chest pain - Cardiac (Cardiac disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (4)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
lightheaded and anxious (General disorders) | 1 (3)
Feeding tube dependency (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Muscle weakness - lower limbs (Musculoskeletal and connective tissue disorders) | 2 (2)
Stupor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (4)
Seroma (Blood and lymphatic system disorders) | 1 (2)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalization - Failure to thrive (General disorders) | 1 (2)
Generalized weakness (General disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Tracheal Hemorrhage (Skin and subcutaneous tissue disorders) | 1 (3)
Wound complication (Surgical and medical procedures) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Paclitaxel, Carboplatin) (N=34)
abnormal electrocardiogram (Cardiac disorders) | 1 (1)
Pain - Abdominal (Gastrointestinal disorders) | 4 (4)
Abodminal distention (Gastrointestinal disorders) | 1 (1)
acid reflux (Gastrointestinal disorders) | 1 (1)
Adrenal insufficiency (Renal and urinary disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Alkaline Phosphatase Increased (Hepatobiliary disorders) | 1 (1)
Allergic reaction (General disorders) | 1 (1)
Alopecia (Immune system disorders) | 18 (18)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Anorexia (Psychiatric disorders) | 8 (8)
Anxiety (Psychiatric disorders) | 6 (6)
Aphonia (General disorders) | 4 (4)
Pain - arm (General disorders) | 3 (3)
Pain - Joint (General disorders) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia - Aspiration (Infections and infestations) | 2 (2)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - back (General disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Pain - bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - chest (General disorders) | 2 (2)
Chest tightness (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Impaired concentration (Nervous system disorders) | 2 (2)
Confusion (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (18)
Cough (General disorders) | 11 (11)
Death (General disorders) | 1 (1)
decreased appetite (Gastrointestinal disorders) | 1 (1)
decreased platelet count (Blood and lymphatic system disorders) | 1 (1)
decreased range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 26 (26)
discomfort (General disorders) | 1 (1)
discomfort - urination & bowel movement (Renal and urinary disorders) | 1 (1)
dizziness (Ear and labyrinth disorders) | 5 (5)
Drooling (General disorders) | 3 (3)
Dry mouth (General disorders) | 6 (6)
epistaxis (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (5)
Dysphagia (General disorders) | 22 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Imbalance (Ear and labyrinth disorders) | 1 (1)
Ear fullness (Ear and labyrinth disorders) | 1 (1)
Pain - ear (Ear and labyrinth disorders) | 3 (3)
edema (Vascular disorders) | 19 (19)
Elevated A1C (Metabolism and nutrition disorders) | 1 (1)
elevated blood cholesterol (Blood and lymphatic system disorders) | 1 (1)
epididymo-orchitis (Reproductive system and breast disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7)
Fatigue (General disorders) | 34 (34)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (Immune system disorders) | 1 (1)
Fibrosis - Deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Influenza-like illness (General disorders) | 4 (4)
Delirium (Nervous system disorders) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Asthenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Granulocytosis (Infections and infestations) | 1 (1)
headache (General disorders) | 6 (6)
Hearing loss (Ear and labyrinth disorders) | 2 (2)
singultus (Gastrointestinal disorders) | 1 (1)
hypothyroidism (Blood and lymphatic system disorders) | 4 (4)
Dysphonia (General disorders) | 9 (9)
Hyperglycemia (Hepatobiliary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypertriglyceridemia (Hepatobiliary disorders) | 1 (1)
hyperkalemia (Blood and lymphatic system disorders) | 2 (2)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
hypotension (Cardiac disorders) | 2 (2)
hypothyroidism (Metabolism and nutrition disorders) | 3 (3)
Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Hypersalivation (Hepatobiliary disorders) | 1 (1)
mucous hypersecretion (Hepatobiliary disorders) | 4 (4)
Cellulitis (Infections and infestations) | 2 (2)
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8)
weakness - lower lip (Musculoskeletal and connective tissue disorders) | 1 (1)
Numbness - neck (Skin and subcutaneous tissue disorders) | 1 (1)
irritation - eyelid (Skin and subcutaneous tissue disorders) | 1 (1)
left auricle keratosis (Cardiac disorders) | 1 (1)
ear fluid drainage (Ear and labyrinth disorders) | 1 (1)
Pain - leg (Musculoskeletal and connective tissue disorders) | 1 (1)
weakness - leg (Musculoskeletal and connective tissue disorders) | 2 (2)
increased libido (Reproductive system and breast disorders) | 1 (1)
Presyncope (Vascular disorders) | 3 (3)
Hyperlipasemia (Hepatobiliary disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Lymphopenia (Immune system disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Otalgia (Ear and labyrinth disorders) | 3 (3)
Halitosis (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Skin and subcutaneous tissue disorders) | 8 (8)
oral mucositis (Skin and subcutaneous tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17)
rhinitis (Infections and infestations) | 2 (2)
necrosis - left lateral intra oral free flap (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 15 (15)
nocturnal hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
oral mucositis (Skin and subcutaneous tissue disorders) | 3 (3)
Pain - oral (General disorders) | 3 (3)
Pain - General (General disorders) | 17 (17)
paresthesia (Skin and subcutaneous tissue disorders) | 13 (13)
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (3)
Platelet count decrease (Blood and lymphatic system disorders) | 9 (9)
Post nasal drip (General disorders) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 3 (3)
Radiation dermatitus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 16 (16)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (General disorders) | 1 (1)
right elbow redness (Skin and subcutaneous tissue disorders) | 1 (1)
Right Foot drop (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1)
Mouth Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 2 (2)
Seroma (Blood and lymphatic system disorders) | 1 (1)
Serum amylase increased (Blood and lymphatic system disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
soft tissue infection (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Pain - Throat (General disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrush (Infections and infestations) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tongue Numbness (General disorders) | 2 (2)
Pain - Tongue (General disorders) | 1 (1)
Tracheal Hemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 3 (3)
Ulceration (Infections and infestations) | 1 (1)
Rash - Upper Chest (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Epiphora (Eye disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight Change (General disorders) | 2 (2)
weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 10 (10)
Wound (Skin and subcutaneous tissue disorders) | 2 (2)
Wound complications (Skin and subcutaneous tissue disorders) | 1 (1)
Wound dehiscence (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03342911/Prot_SAP_000.pdf